CLINICAL TRIAL: NCT00812162
Title: Effects of Dietary Pork and Egg on Appetite, Meal-patterning, and Weight Loss in Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Wayne Campbell, Ph.D., Purdue University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0610004602; Pork Board 1320067860 (Other: National Pork Board); Egg Board 1320067903 (Other: American Egg Board)
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): High protein diet.
  Interventions: Other: Energy Restriction
- 2 (Experimental): Lower protein diet.
  Interventions: Other: Energy Restriction

INTERVENTIONS:
Other: Energy Restriction — Energy restricted diet of 750 kcal less than subjects requirement with a high protein diet.
  Arms: 1
Other: Energy Restriction — Energy restricted diet of 750 kcal less than subjects requirement with a lower protein diet.
  Arms: 2

SUMMARY:
The purpose of this study is to identify how adult men respond to a weight loss diet that includes pork and eggs and increasing the number of meals consumed throughout the day. This is a 13-week study (12-weeks of weight loss and 1-week of baseline measurement).

ELIGIBILITY:
Inclusion Criteria:

* Age range: 21 years and older
* Body mass index between 25.0-39.9 kg/m2
* Weight stable (< 4.5 kg (~10 lbs) weight gain or loss within last 6 months)
* Body fat >25% (assessed by skinfold and plethysmography (if needed))
* Non-smoking (within the last 6 months)
* Constant habitual activity patterns (within last 3 months)
* Clinically normal blood profiles (specifically, normal liver and kidney function; fasting blood glucose <110 mg/dl)
* Not taking medications known to influence appetite or metabolism
* Non-diabetic

Exclusion Criteria:

* Age: <21 years
* Body mass index: outside of the 25.0-39.9 kg/m2 range
* Gained or lost > 4.5 kg (10 lbs) within the last 6 months
* Body fat <25% as assessed by plethysmography
* Smoker (currently or within the last 6 months)
* Intermittently been involved in a diet and/or exercise program within the last 3 months
* Clinically abnormal blood profiles as identified by our study physician, Arthur Rosen, MD
* Taking medications (currently or within the last 3 months) known to influence appetite or metabolism
* Clinically diagnosed as diabetic
* Allergies to eggs
* Lactose intolerance
* Clinically diagnosed with diverticulosis
* Clinically diagnosed with diverticulitis

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-01; Primary Completion 2009-02 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The primary aim is to examine the effects of increased protein intake on appetite, selected appetite hormones (insulin, leptin, ghrelin), whole body energy expenditure, and body composition (fat mass and fat-free mass) changes. | 12 week

SECONDARY OUTCOMES:
The secondary aim of this study is to evaluate the effects of meal frequency on appetite by asking the men to frequently rate their appetite on days that they purposefully eat 3 vs. 6 times/day. | 12 week

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Campbell, Ph.D., Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States